CLINICAL TRIAL: NCT05035485
Title: Maternal Cardiac Output Response to Rescue Norepinephrine and Phenylephrine Boluses During Spinal Anesthesia for Caesarean Section in Patients With Severe Preeclampsia: a Randomized, Controlled Trial
Brief Title: Maternal Cardiac Output Response to Rescue Norepinephrine and Phenylephrine Boluses in Patients With Severe Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2021-2
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Hemodynamic Instability
Keywords: Cardiac output response; Norepinephrine; Phenylephrine; Preeclampsia; Cesarean section
MeSH Terms: conditions — Pre-Eclampsia | interventions — Phenylephrine; Vasoconstrictor Agents; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenylephrine group (Active Comparator): Rescue phenylephrine (75μg) was given when postspinal anesthesia hypotension occurred
  Interventions: Drug: Phenylephrine
- Norepinephrine group (Experimental): Rescue norepinephrine (6μg) was given when postspinal anesthesia hypotension occurred
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Phenylephrine — A rescue phenylephrine (75μg) was given when postspinal anesthesia hypotension occurred within 30 minutes after spinal anesthesia
  Other Names: Vasopressors
  Arms: Phenylephrine group
Drug: Norepinephrine — A rescue norepinephrine (6μg) was given when postspinal anesthesia hypotension occurred within 30 minutes after spinal anesthesia
  Other Names: Vasopressors
  Arms: Norepinephrine group

SUMMARY:
The purpose of this study is to investigate the maternal cardiac output response to rescue norepinephrine and phenylephrine boluses for postspinal anesthesia hypotension in parturients with preeclampsia undergoing cesarean section.

DETAILED DESCRIPTION:
Preeclampsia, which affects 5% to 7% of parturients, is a significant cause of maternal and neonatal morbidity and mortality. Because of constricted myometrial spiral arteries with exaggerated vasomotor responsiveness, though blood pressure in parturients with preeclampsia are apparently higher than healthy parturients, placental hypoperfusion is more common. Spinal anesthesia is still the preferred mode of anesthesia in parturients with preeclampsia for cesarean section. In preeclampsia parturients, spinal anesthesia improve intervillous blood flow (provided that hypotension is avoided) which contribute to increase placental perfusion. Even so, 17-26% parturients with preeclampsia experienced postspinal anesthesia hypotension due to the extensive sympathetic block that occurred with spinal anesthesia. As a potential substitute drug for phenylephrine and ephedrine, norepinephrine has gained traction for use in parturients undergoing cesarean section. However, hemodynamic effects of the rescue norepinephrine bolus is still unknown. The purpose of this study is to investigate the maternal cardiac output response to rescue norepinephrine and phenylephrine boluses for postspinal anesthesia hypotension in parturients with preeclampsia undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Primipara or multipara
* Singleton pregnancy ≥32 weeks
* American Society of Anesthesiologists physical status classification II to III
* Scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Baseline blood pressure ≥180 mmHg
* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-01-21 (Actual)

PRIMARY OUTCOMES:
Cardiac output (CO) | 1-30 minutes after spinal anesthesia.
  Evaluated by the VIGILCO monitoring system.
Stroke volume (SV) | 1-30 minutes after spinal anesthesia
  Evaluated by the VIGILCO monitoring system.
Systemic vascular resistance (SVR) | 1-30 minutes after spinal anesthesia
  Evaluated by the VIGILCO monitoring system.

SECONDARY OUTCOMES:
Overall stability of systolic blood pressure control versus baseline | 1-30 minutes after spinal anesthesia
  Evaluated by performance error (PE)
Overall stability of heart rate control versus baseline | 1-30 minutes after spinal anesthesia
  Evaluated by performance error (PE)
The incidence of post-spinal anesthesia hypotension | 1-30 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension. | 1-30 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) < 60% of the baseline
The incidence of nausea and vomiting. | 1-30 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of bradycardia. | 1-30 minutes after spinal anesthesia
  Heart rate < 60 beats/min.
The incidence of hypertension. | 1-30 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline.
pH | Immediately after delivery
  From umbilical arterial blood gases.
Partial pressure of oxygen (PO2) | Immediately after delivery
  From umbilical arterial blood gases.
Base excess (BE) | Immediately after delivery
  From umbilical arterial blood gases.
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Study Chair — General Hospital of Ningxia Medical University; Xiangzhao Xu, M.D.; Ph. D, Study Chair — The People's Hospital of Nanchuan
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China